CLINICAL TRIAL: NCT03562377
Title: A Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Effect of Tralokinumab on Vaccine Antibody Responses in Adults With Moderate-to-severe Atopic Dermatitis Who Are Candidates for Systemic Therapy
Brief Title: Vaccine Responses in Tralokinumab-Treated Atopic Dermatitis - ECZTRA 5 (ECZema TRAlokinumab Trial No. 5)
Acronym: ECZTRA 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-1341
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor any of the investigator or LEO staff who are involved in the treatment or clinical evaluation and monitoring of the subjects will be aware of the treatment received. The packaging and labelling of tralokinumab/placebo will contain no evidence of their identity.
  Since tralokinumab and placebo are visually distinct and not matched for viscosity, they will be handled and administered by a qualified, unblinded healthcare professional at the trial site who will not be involved in the management of trial subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tralokinumab (Experimental): Week 0 to 16:
  Tralokinumab will be given as subcutaneous injections.
  Subjects will receive a tralokinumab loading dose at Day 0 followed by tralokinumab injection regimen A. The last administration will occur at Week 14.
  Interventions: Drug: Tralokinumab; Biological: Tdap vaccine; Biological: Meningococcal vaccine
- Placebo (Placebo Comparator): Placebo (dummy treatment) will be given as subcutaneous injections.
  Subjects will receive a placebo loading dose at Day 0 followed by placebo injection regimen A. The last administration will occur at Week 14.
  Interventions: Drug: Placebo; Biological: Tdap vaccine; Biological: Meningococcal vaccine

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous administration.
  Arms: Tralokinumab
Drug: Placebo — Placebo contains the same excipients in the same concentration only lacking tralokinumab.
  Arms: Placebo
Biological: Tdap vaccine — Tetanus (lockjaw), diphtheria (infection of the nose and throat), and pertussis (whooping cough) vaccine. All subjects will receive 1 dose at Week 12.
Biological: Meningococcal vaccine — This vaccine is used to prevent meningococcal diseases (infection of the brain and spinal cord) and blood poisoning. All subjects will receive 1 dose at Week 12.

SUMMARY:
The purpose of this trial is to test if treatment with the trial drug, tralokinumab, can affect the body's immune response to vaccines. The trial will also evaluate the efficacy of tralokinumab when it is given concomitantly with vaccines.

The trial includes a screening period of 2 to 6 weeks, a treatment period of 16 weeks (Weeks 0 to 16), and a 14-week off-treatment follow-up period for the assessment of safety (Weeks 16 to 30). Eligible subjects may transfer to an open-label, long-term trial at Week 16 or later.

DETAILED DESCRIPTION:
Subjects with atopic dermatitis (AD) will be treated with either tralokinumab or dummy treatment (placebo) for 16 weeks. All subjects will receive 2 vaccines at Week 12. The vaccines are:

1. Tetanus (lockjaw), diphtheria (infection of the nose and throat), and pertussis (whooping cough) vaccine. This combination vaccine is also known as the Tdap vaccine and is used to prevent these 3 diseases.
2. Meningococcal vaccine. This vaccine is used to prevent meningococcal diseases (infection of the brain and spinal cord) and blood poisoning.

The primary objective of the trial is to demonstrate non-inferiority of tralokinumab versus placebo with respect to immune responses to concomitantly administered vaccines.

The secondary objective is to evaluate efficacy of tralokinumab concomitantly administered with vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 54 years
* Diagnosis of AD as defined by Hanifin and Rajka (1980) criteria for AD
* History of AD for ≥1 year
* Subjects who have a recent history of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable
* AD involvement of ≥10% body surface area at screening and baseline
* An EASI score of ≥12 at screening and 16 at baseline
* An IGA score of ≥3 at screening and at baseline
* Subjects must have applied a stable dose of emollient twice daily (or more, as needed) for at least 14 days before randomisation

Exclusion Criteria:

* Subjects for whom administration of the meningococcal vaccine provided in this trial is contraindicated or medically inadvisable, according to local label of the vaccine
* Subjects for whom administration of the tetanus, diphtheria, and pertussis vaccine provided in this trial is contraindicated or medically inadvisable, according to local label of the vaccine
* Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment
* Use of tanning beds or phototherapy within 6 weeks prior to randomization
* Treatment with systemic immunosuppressive/immunomodulating medications and/or systemic corticosteroids within 4 weeks prior to randomization
* Treatment with the topical medications topical corticosteroids (TCS), topical calcineurin inhibitor (TCI) or phosphodiesterase 4 (PDE-4) inhibitor within 2 weeks prior to randomization
* Receipt of any vaccine (except influenza virus vaccines) within 3 months prior to screening, any meningococcal vaccine within 1 year prior to screening, or any tetanus-, diphtheria-, or pertussis-containing vaccine within 5 years prior to screening
* Receipt of any marketed (i.e. immunoglobulin, anti-IgE) or investigational biologic agent, including dupilumab
* History of any active skin infection within 1 week prior to randomization
* History of a clinically significant infection (systemic infection or serious skin infection requiring parenteral treatment) within 4 weeks prior to randomization

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (48):
- United States (37):
  - Leo Pharma Investigational Site, Fort Smith, Arkansas
  - LEO Pharma Investigational Site, Bakersfield, California
  - Leo Pharma Investigational Site, Beverly Hills, California
  - Leo Pharma Investigational Site, Fountain Valley, California
  - Leo Pharma Investigational Site, Los Angeles, California
  - Leo Pharma Investigational Site, Newport Beach, California
  - LEO Pharma Investigational Site, San Diego, California
  - LEO Pharma Investigational Site, Centennial, Colorado
  - LEO Pharma Investigational Site, Denver, Colorado
  - LEO Pharma Investigational Site, Thornton, Colorado
  - Leo Pharma Investigational Site, Coral Gables, Florida
  - Leo Pharma Investigational Site, Doral, Florida
  - Leo Pharma Investigational Site, Hialeah, Florida
  - LEO Pharma Investigational Site, Atlanta, Georgia
  - Leo Pharma Investigational Site, New Albany, Indiana
  - Leo Pharma Investigational Site, South Bend, Indiana
  - LEO Pharma Investigational Site, Bangor, Maine
  - Leo Pharma Investigational Site, Boston, Massachusetts
  - LEO Pharma Investigational Site, Brighton, Massachusetts
  - Leo Pharma Investigational Site, Ann Arbor, Michigan
  - LEO Pharma Investigational Site, Southfield, Michigan
  - Leo Pharma Investigational Site, Missoula, Montana
  - Leo Pharma Investigational Site, East Windsor, New Jersey
  - LEO Pharma Investigational Site, Brooklyn, New York
  - Leo Pharma Investigational Site, Cortland, New York
  - Leo Pharma Investigational Site, Forest Hills, New York
  - Leo Pharma Investigational Site, New York, New York
  - Leo Pharma Investigational Site, Cincinnati, Ohio
  - LEO Pharma Investigational Site, Cincinnati, Ohio
  - LEO Pharma Investigational Site, Gahanna, Ohio
  - LEO Pharma Investigational Site, Medford, Oregon
  - Leo Pharma Investigational Site, Chattanooga, Tennessee
  - Leo Pharma Investigational Site, Austin, Texas
  - LEO Pharma Investigational Site, Dallas, Texas
  - Leo Pharma Investigational Site, Frisco, Texas
  - Leo Pharma Investigational Site, South Burlington, Vermont
  - Leo Pharma Investigational Site, Spokane, Washington
- Canada (11):
  - LEO Pharma Investigational Site, Edmonton, Alberta
  - LEO Pharma Investigational Site, Vancouver, British Colombia
  - LEO Pharma Investigational Site, St. John's, Newfoundland and Labrador
  - LEO Pharma Investigational Site, Hamilton, Ontario
  - LEO Pharma Investigational Site, London, Ontario
  - LEO Pharma Investigational Site, Oakville, Ontario
  - LEO Pharma Investigational Site, Peterborough, Ontario
  - LEO Pharma Investigational Site, Richmond Hill, Ontario
  - LEO Pharma Investigational Site, Toronto, Ontario
  - LEO Pharma Investigational Site, Windsor, Ontario
  - LEO Pharma Investigational Site, Verdun, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tralokinumab: Participants received tralokinumab every 2 weeks for 16 weeks, and the Tdap and meningococcal vaccines at Week 12.
- Placebo: Participants received placebo every 2 weeks for 16 weeks, and the Tdap and meningococcal vaccines at Week 12.
Period: Treatment Period
Arm/Group | Tralokinumab | Placebo
Started | 107 (Number of participants assigned to treatment) | 108 (Number of participants assigned to treatment)
Safety Analysis Set (Defined as all participants randomised to treatment who were exposed to IMP (tralokinumab/placebo).) | 107 | 107
Per Protocol Anaysis Set (Excluding participants who did not receive vaccines, violated selected eligiblity criteria, etc.) | 88 | 78
Full Analysis Set (Defined as all participants randomised to treatment who were exposed to IMP (tralokinumab/placebo)) | 106 | 108
Completed | 100 (Number of participants attending the Week 16 visit (end of treatment visit)) | 89 (Number of participants attending the Week 16 visit (end of treatment visit))
Not Completed | 7 | 19
Period: Safety Follow-up Period
Arm/Group | Tralokinumab | Placebo
Started | 75 (Last contact after exposure end. Main reason for not entering follow-up: transfer to extension trial) | 75 (Last contact after exposure end. Main reason for not entering follow-up: transfer to extension trial)
Completed | 16 (Attended Week 30 visit. Main reason for not attending was transfer to long-term extension trial.) | 18 (Attended Week 30 visit. Main reason for not attending was transfer to long-term extension trial.)
Not Completed | 59 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tralokinumab | Placebo | Total
Number analyzed (Participants) | 107 | 108 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 108 | 215
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (11.2) | 34.4 (10.8) | 34.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 73 | 126
  Male | 54 | 35 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 19 | 36
  Not Hispanic or Latino | 90 | 89 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 18 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 25 | 27 | 52
  White | 62 | 56 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 35 | 69
  United States | 73 | 73 | 146
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — The IGA is an instrument used in clinical trials to rate the severity of the subject's global atopic dermatitis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    Clear (IGA=0) | 0 | 0 | 0
    Almost clear (IGA=1) | 0 | 0 | 0
    Mild disease (IGA=2) | 0 | 0 | 0
    Moderate disease (IGA=3) | 72 | 72 | 144
    Severe disease (IGA=4) | 34 | 36 | 70
    Missing | 1 | 0 | 1
Eczema Area and Severity Index score [Mean (Standard Deviation); unit: units on a scale] — The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
  units on a scale | 26.26 (10.79) | 26.75 (11.23) | 26.51 (11.00)

OUTCOME MEASURES:

1. Primary Outcome: Positive Anti-tetanus Response at Week 16
Description: The antibody response to Tdap vaccine will be assessed by measuring serum anti-tetanus IgG by an immunoassay. A positive response is defined as a 3-fold IgG increase compared to Week 12 if IgG ≤1.0 IU/mL at Week 12; or IgG ≥2.5 IU/mL if IgG >1.0 IU/mL at Week 12.
Time Frame: Week 12 to Week 16
Population: The per protocol analysis set was used for the primary analysis, excluding participants who did not provide vaccine response data at Week 12 (1 participant in the tralokinumab group and 2 participants in the placebo group).
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 87 | 76
Participants | 80 | 73
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Non-Inferiority — The difference in response rates was calculated using the Mantel-Haenszel estimate of the risk difference stratified by baseline disease severity together with the 2-sided 95% CI. Non-inferiority of tralokinumab was demonstrated if the lower limit of the 95% CI was greater than -25%. Power calculation assumed 160 subjects in the per protocol analysis set, providing 98% power to establish non-inferiority, assuming response rates of 80% in both treatment groups and a non-inferiority margin of -25%; Mantel Haenszel; Risk Difference (RD) = -4.1, 95% CI 2-sided [-11.3 to 3.1]

2. Primary Outcome: Positive Anti-meningococcal Response at Week 16
Description: The antibody response to meningococcal vaccine will be assessed by measuring serum anti-meningococcal IgG by an immunoassay. A positive response is defined as at least a 3-fold increase compared to Week 12.
Time Frame: Week 12 to Week 16
Population: The per protocol analysis set was used for the primary analysis, excluding participants who did not provide vaccine response data at Week 12 (2 participants in each treatment group).
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 86 | 76
Participants | 74 | 64
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mantel Haenszel; Risk Difference (RD) = 1.8, 95% CI 2-sided [-9.2 to 12.8]

3. Secondary Outcome: Participants With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: The IGA is an instrument used in clinical trials to rate the severity of the subject's global atopic dermatitis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Week 0 to Week 16
Population: The analysis of the secondary outcome measures was done for the full analysis set, i.e. all subjects who were randomised and exposed to IMP (tralokinumab/placebo). 1 subject in the tralokinumab group was randomised in error and not exposed to IMP and therefore excluded from the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 106 | 108
Participants | 33 | 21
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel — The p-value was adjusted for multiplicity by a pre-specified testing hierarchy. Subjects with missing data or subjects who received rescue medication prior to Week 16 were considered non-responders in the primary analysis of the primary estimand; The difference in response rates was analysed using the Cochran-Mantel-Haenszel test stratified by baseline disease severity (moderate or severe); Risk Difference (RD) = 11.4, 95% CI 2-sided [0.2 to 22.6]

4. Secondary Outcome: Participants Achieving at Least 75% Reduction in Eczema Area and Severity Index (EASI) at Week 16.
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis.
  > The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Time Frame: Week 0 to Week 16
Population: The analysis of the secondary outcome measures was done for the full analysis set, i.e. all participants who were randomised and exposed to IMP (tralokinumab/placebo). 1 participant in the tralokinumab group was randomised in error and not exposed to IMP and therefore excluded from the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 106 | 108
Participants | 52 | 39
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Test type: Superiority; p = 0.057, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Risk Difference (RD) = 12.7, 95% CI 2-sided [-0.2 to 25.7]

5. Secondary Outcome: Number of AEs.
Description: Overall summary of AEs during the treatment period is presented. For list of SAEs and frequent AEs by MedDRA system organ class (SOC) and preferred term (PT) during the entire trial period (including safety follow-up), see Adverse Events Overview section.
Time Frame: Week 0 to Week 16
Population: The descriptive analysis was performed on the safety analysis set. The safety analysis set was defined as all participants who received at least 1 dose of IMP during the trial. Subjects who received at least 1 dose of tralokinumab were analysed in the tralokinumab group.
Measure: Number; unit: AEs
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 107 | 107
AEs | 112 | 133

6. Secondary Outcome: Presence of Anti-drug Antibodies (ADA).
Description: ADA levels were measured using a validated bioanalytical method. Data were reported in the following categories: positive (presence of ADA at baseline and/or presence of ADA at at least 1 post-baseline assessment), perishing (presence of ADA at baseline and absence of ADA at all post-baseline assessments), negative (absence of ADA at all assessments), no post-baseline ADA assessment.
Time Frame: Week 0 to Week 16
Population: All subjects in the safety analysis set were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 107 | 107
Participants
  Positive | 2 | 4
  Perishing | 1 | 2
  Negative | 103 | 97
  No post-baseline ADA assessment | 1 | 4

ADVERSE EVENTS:
Time Frame: AEs were collected from time of first trial-related activity after the subject had signed the ICF until completion of the clinical trial (defined as the safety follow up visit at Week 30). Non-serious AEs possibly/probably related to IMP and ongoing at the time of trial completion were followed up for 2 weeks or until final outcome, whichever came first. Serious AEs were followed up until final outcome had been established.
Groups:
- Tralokinumab: Tralokinumab
- Placebo: Placebo
Arm/Group | Tralokinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 3/107 | 3/107
Other Adverse Events (participants affected / at risk) | 27/107 | 25/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab (N=107) | Placebo (N=107)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab (N=107) | Placebo (N=107)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Seasonal allergy (Immune system disorders) | 3 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (7)
Viral upper respiratory tract infection (Infections and infestations) | 10 (10) | 3 (4)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 12 (14) | 13 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all phase 3 clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT03562377/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03562377/SAP_001.pdf